CLINICAL TRIAL: NCT05740735
Title: Emotional and Neutral Sounds for Neurophysiological Prognostic Assessment of Critically Ill Patients With a Disorder of Consciousness (DOC)
Brief Title: Emotional and Neutral Sounds for Neurophysiological Prognostic Assessment of Critically Ill Patients With a Disorder of Consciousness
Acronym: ExpressComa
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220568; 2022-A00607-36 (Other: France : ANSM)
Record Dates: First submitted 2022-09-06; First posted 2023-02-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Disorder of Consciousness
Keywords: Disorder of consciousness; Cardiac arrest; Coma; Intensive care unit; Neuro-prognostication; Event related potential (ERP); Electroencephalogram (EEG); Emotional sounds; Subject own name (SON); P300; Mismatch negativity (MMN)
MeSH Terms: conditions — Consciousness Disorders; Heart Arrest; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Disorder of consciousness patients - Prospective group: DOC defined either by a coma (Glasgow Coma Scale <8), a vegetative state (VS) or a minimal state of consciousness (MCS) according to the Coma recovery scale-revised (CRS-r) after a primary brain injury: severe traumatic brain injury (TBI)), subarachnoid hemorrhage, stroke or cardiac arrest (CA)
  Interventions: Other: Use of "expressive" sounds
- Disorder of consciousness patients - Retrospective group
  Interventions: Other: Having benefited from a prognostic evaluation by event related potentials (without sound research methods, only neutral sounds)

INTERVENTIONS:
Other: Use of "expressive" sounds — Use of "expressive" sounds, that is to say the own first name pronounced by the voice of the relative to generate the P300 and a sound with an "approaching" character of the subject to generate the MMN.
  The investigators will thus be able to compare:
  * MMN: present/absent for each modality (neutral vs approaching sounds)
  * Wave P3a: latencies and amplitudes for each modality (own first name voice of the near vs unfamiliar).
  Groups: Disorder of consciousness patients - Prospective group
Other: Having benefited from a prognostic evaluation by event related potentials (without sound research methods, only neutral sounds) — Retrospective inclusion Have already had an assessment with event related potentials without "emotional" modalities (VF and similar sounds) as part of their care between April 2022 and December 2022 in intensive care at Cochin hospital.
  Groups: Disorder of consciousness patients - Retrospective group

SUMMARY:
The purpose of this study is to determine if the use of emotional sound as subject own name (SON) pronounced by a familiar voice (FV) compared to SON pronounced by a non-familiar voice (NFV) during event related potential (ERP) produced a more reliable neurophysiological P300 responses, and to assess the prognostic value of this P300 responses induced by the SON with a FV.

DETAILED DESCRIPTION:
The evaluation of the neurological outcome of intensive care unit (ICU) patients with a disorder of consciousness (DOC) is a major medical, ethical and economic issue. These DOC are essentially related to a direct anoxo-ischaemic (post-cardiac arrest), traumatic or even vascular (caused by a hemorrhagic or ischemic vascular accident) cerebral aggression. The techniques currently available, whether neurophysiological (electroencephalogram (EEG) and evoked potentials (EP)), neuroradiological or biological, only allow an approximate evaluation for a large number of aetiologies and patients (Obadi. EEG and EPs have the advantage of being feasible at the patient's bedside, with a precise spatial-temporal resolution of the cerebral capacities to integrate sensory stimulation. If some neurophysiological tests have an imperfect predictive capacity, event-related potentials, (ERPs) with "oddball paradigm" seem to be a promising method. During their realizations by exposing the subject to listening to a deviant and rare auditory stimulus within other frequent stimuli, a first neurophysiological response is generated 150 to 200ms after the stimulation called "mismatch negativity" (MMN), then a second response to 300ms of stimulation called "P3a" is generated. The latter would reflect the orientation of a subject's attention towards the deviant stimulus and could predict arousal.

Some recent data report that a P3 response obtained by exposing the subject to a stimulus with expressive and emotional value, such as the patient's own first name, could improve the prognostic value of this neurophysiological tool (Fischer et al, Holeckova et al). Indeed, the neural processing of expressive voices involves a greater number of subcortical and cortical regions than neutral sounds (Schirmer and Kotz). Moreover, some data suggest that the use of a "subject own name" (SON) auditory stimulus pronounced by a familiar voice (FV) compared to an unfamiliar voice (NFV) could improve the prognostic value of P3 or even the use binaural sounds with a three-dimensional effect as "looming" or "receding" sounds, these hypotheses having never been evaluated in DOC patients.

The investigators hypothesize that cortical and subcortical activation is more complex and intense in response to emotional than to neutral sounds, and that obtaining a P3a response generated by sounds expressive type SON pronounced by a familiar voice (FV) would have a prognostic value greater than the P3 response induced by the SON with an unfamiliar voice for wakefulness prediction of DOC patients; The investigators will also test the hypothesis that the prognostic value of the MMN response generated by sounds with randomly varied motion in their 3D auditory field (e.g. looming or receding sources) is higher than those generated by neutral sounds.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in ICU for cardiac arrest, stroke, subarachnoid haemorrhage or head trauma,
* persistent disorder of consciousness (DoC) 12 hours after sedation weaning or patient who has benefited from a prognostic assessment for persistent DoC and who has had in this assessment an evaluation by late PEA with MMN and P300 responses only to neutral sounds ("beep" and patient's first name pronounced by an unfamiliar voice) there is more than 6 months (since April 2022)

Exclusion Criteria:

* Moribund patient
* Uncontrolled Shock during the neurophysiological evaluation
* Sedated patient
* Minor patient
* brain death
* Known deafness
* Pregnant woman
* Prior inclusion in the study
* Patient not affiliated to a social security system
* Implementation of limitations and stop of active therapies
* Patient under legal protection
* Patient benefiting from State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Cochin Hospital ICU with a primary brain injury (after CA, TBI, stroke) and a persistent DOC (coma, VS, MCS) 12 hours after sedation discontinuation.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | Month 3
  Neurological outcome - From 1 to 8 : 8 = Good Recovery - higher level / 7 = Good Recovery - lower level / 6 = Moderate disability - higher level / 5 = Moderate disability - lower level / 4 = Severe disability - higher level / 3 l= Severe disability - lower level / 2 = Persistent vegetative state / 1 = Death

SECONDARY OUTCOMES:
Glasgow coma scale (GCS) | Day 7
  Level of awareness - From 3 to 15 : Score of 3 to 8 defined comatose state, score 9 to 14 defined alteration of awareness or confusion and score 15 defined conscious and not confuse patients
Glasgow coma scale (GCS) | Day 14
  Level of awareness - From 3 to 15 : Score of 3 to 8 defined comatose state, score 9 to 14 defined alteration of awareness or confusion and score 15 defined conscious and not confuse patients
Richmond Agitation-Sedation Scale | Day 7
  Level of awareness - From -5 to + 4 : +4 = Combative Overtly combative, violent, immediate danger to staff / +3 = Very agitated Pulls or removes tube(s) or catheter(s); aggressive / +2 = Agitated Frequent non-purposeful movement, fights ventilator / +1 = Restless Anxious but movements not aggressive vigorous / 0 = Alert and calm / -1 = Drowsy Not fully alert, but has sustained awakening / (eye-opening/eye contact) to voice (>10 seconds) / -2 = Light sedation Briefly awakens with eye contact to voice (<10 seconds) / -3 = Moderate sedation Movement or eye opening to voice (but no eye contact) / -4 = Deep sedation No response to voice, but movement or eye opening to physical stimulation / -5 = Unarousable
Richmond Agitation-Sedation Scale | Day 14
  Level of awareness - From -5 to + 4 : +4 = Combative Overtly combative, violent, immediate danger to staff / +3 = Very agitated Pulls or removes tube(s) or catheter(s); aggressive / +2 = Agitated Frequent non-purposeful movement, fights ventilator / +1 = Restless Anxious but movements not aggressive vigorous / 0 = Alert and calm / -1 = Drowsy Not fully alert, but has sustained awakening / (eye-opening/eye contact) to voice (>10 seconds) / -2 = Light sedation Briefly awakens with eye contact to voice (<10 seconds) / -3 = Moderate sedation Movement or eye opening to voice (but no eye contact) / -4 = Deep sedation No response to voice, but movement or eye opening to physical stimulation / -5 = Unarousable
Coma recovery scale-revised CRS-r | Day 7
  Level of awareness - From 0 to 23 : 0 to 7 = vegetative state, 8 to 15 = minimal conscious state, 16-23 = minimal conscious state emergence
Coma recovery scale-revised CRS-r | Day 14
  Level of awareness - From 0 to 23 : 0 to 7 = vegetative state, 8 to 15 = minimal conscious state, 16-23 = minimal conscious state emergence
Glasgow Outcome Scale-Extended (GOS-E) | Day 28
  Neurological outcome - From 1 to 8 : 8 = Good Recovery - higher level / 7 = Good Recovery - lower level / 6 = Moderate disability - higher level / 5 = Moderate disability - lower level / 4 = Severe disability - higher level / 3 l= Severe disability - lower level / 2 = Persistent vegetative state / 1 = Death
Glasgow Outcome Scale-Extended (GOS-E) | Intensive care unit discharge, up to 6 months
  Neurological outcome - From 1 to 8 : 8 = Good Recovery - higher level / 7 = Good Recovery - lower level / 6 = Moderate disability - higher level / 5 = Moderate disability - lower level / 4 = Severe disability - higher level / 3 l= Severe disability - lower level / 2 = Persistent vegetative state / 1 = Death
Richmond Agitation-Sedation Scale | Day 28
  Neurological outcome - From -5 to + 4 : +4 = Combative Overtly combative, violent, immediate danger to staff / +3 = Very agitated Pulls or removes tube(s) or catheter(s); aggressive / +2 = Agitated Frequent non-purposeful movement, fights ventilator / +1 = Restless Anxious but movements not aggressive vigorous / 0 = Alert and calm / -1 = Drowsy Not fully alert, but has sustained awakening / (eye-opening/eye contact) to voice (>10 seconds) / -2 = Light sedation Briefly awakens with eye contact to voice (<10 seconds) / -3 = Moderate sedation Movement or eye opening to voice (but no eye contact) / -4 = Deep sedation No response to voice, but movement or eye opening to physical stimulation / -5 = Unarousable
Richmond Agitation-Sedation Scale | Intensive care unit discharge, up to 6 months
  Neurological outcome - From -5 to + 4 : +4 = Combative Overtly combative, violent, immediate danger to staff / +3 = Very agitated Pulls or removes tube(s) or catheter(s); aggressive / +2 = Agitated Frequent non-purposeful movement, fights ventilator / +1 = Restless Anxious but movements not aggressive vigorous / 0 = Alert and calm / -1 = Drowsy Not fully alert, but has sustained awakening / (eye-opening/eye contact) to voice (>10 seconds) / -2 = Light sedation Briefly awakens with eye contact to voice (<10 seconds) / -3 = Moderate sedation Movement or eye opening to voice (but no eye contact) / -4 = Deep sedation No response to voice, but movement or eye opening to physical stimulation / -5 = Unarousable
Coma recovery scale-revised CRS-r | Day 28
  Neurological outcome - From 0 to 23 : 0 to 7 = vegetative state, 8 to 15 = minimal conscious state, 16-23 = minimal conscious state emergence
Coma recovery scale-revised CRS-r | Intensive care unit discharge, up to 6 months
  Neurological outcome - From 0 to 23 : 0 to 7 = vegetative state, 8 to 15 = minimal conscious state, 16-23 = minimal conscious state emergence
Glasgow Outcome Scale-Extended (GOS-E) | Month 6
  Neurological outcome - From 1 to 8 : 8 = Good Recovery - higher level / 7 = Good Recovery - lower level / 6 = Moderate disability - higher level / 5 = Moderate disability - lower level / 4 = Severe disability - higher level / 3 l= Severe disability - lower level / 2 = Persistent vegetative state / 1 = Death
Mortality | Day 28
Mortality | Month 3
P3a amplitudes responses | At inclusion
  Neurophysiological characteristics of the P3a response to different stimuli (FV vs NFV) / Comparison of the P3a amplitudes and latencies responses according to the different stimuli
P3a latencies responses | At inclusion
  Neurophysiological characteristics of the P3a response to different stimuli (FV vs NFV) / Comparison of the P3a amplitudes and latencies responses according to the different stimuli
MMN amplitudes responses | At inclusion
  Neurophysiological characteristics of the MMN response to the different stimuli (looming or receding sources) / Comparison of the MMN amplitudes and latencies responses according to the different stimuli
MMN latencies responses | At inclusion
  Neurophysiological characteristics of the MMN response to the different stimuli (looming or receding sources) / Comparison of the MMN amplitudes and latencies responses according to the different stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Benghanem, MD, MSc, PhD student, Principal Investigator — Medical ICU Cochin Hospital, APHP.Centre; Alain Cariou, MD, PhD, Study Director — Medical ICU, Cochin Hospital, APHP.Centre
Locations (2):
- France (2):
  - Medical ICU, HEGP Hospital, APHP.Centre, Paris, IDF
  - Medical ICU, Cochin Hospital, APHP.Centre, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre-Obadia N, Zyss J, Gavaret M, Lefaucheur JP, Azabou E, Boulogne S, Guerit JM, McGonigal A, Merle P, Mutschler V, Naccache L, Sabourdy C, Trebuchon A, Tyvaert L, Vercueil L, Rohaut B, Delval A. Recommendations for the use of electroencephalography and evoked potentials in comatose patients. Neurophysiol Clin. 2018 Jun;48(3):143-169. doi: 10.1016/j.neucli.2018.05.038. Epub 2018 May 18. PMID 29784540
- [Background] Comanducci A, Boly M, Claassen J, De Lucia M, Gibson RM, Juan E, Laureys S, Naccache L, Owen AM, Rosanova M, Rossetti AO, Schnakers C, Sitt JD, Schiff ND, Massimini M. Clinical and advanced neurophysiology in the prognostic and diagnostic evaluation of disorders of consciousness: review of an IFCN-endorsed expert group. Clin Neurophysiol. 2020 Nov;131(11):2736-2765. doi: 10.1016/j.clinph.2020.07.015. Epub 2020 Aug 14. PMID 32917521
- [Background] Fischer C, Dailler F, Morlet D. Novelty P3 elicited by the subject's own name in comatose patients. Clin Neurophysiol. 2008 Oct;119(10):2224-30. doi: 10.1016/j.clinph.2008.03.035. Epub 2008 Aug 28. PMID 18760663
- [Background] O'Mahony D, Rowan M, Walsh JB, Coakley D. P300 as a predictor of recovery from coma. Lancet. 1990 Nov 17;336(8725):1265-6. doi: 10.1016/0140-6736(90)92887-n. No abstract available. PMID 1978111
- [Background] Holeckova I, Fischer C, Morlet D, Delpuech C, Costes N, Mauguiere F. Subject's own name as a novel in a MMN design: a combined ERP and PET study. Brain Res. 2008 Jan 16;1189:152-65. doi: 10.1016/j.brainres.2007.10.091. Epub 2007 Nov 12. PMID 18053971
- [Background] Holeckova I, Fischer C, Giard MH, Delpuech C, Morlet D. Brain responses to a subject's own name uttered by a familiar voice. Brain Res. 2006 Apr 12;1082(1):142-52. doi: 10.1016/j.brainres.2006.01.089. PMID 16703673
- [Background] Naccache L, Puybasset L, Gaillard R, Serve E, Willer JC. Auditory mismatch negativity is a good predictor of awakening in comatose patients: a fast and reliable procedure. Clin Neurophysiol. 2005 Apr;116(4):988-9. doi: 10.1016/j.clinph.2004.10.009. Epub 2004 Dec 10. No abstract available. PMID 15792909
- [Background] Liegeois-Chauvel C, Benar C, Krieg J, Delbe C, Chauvel P, Giusiano B, Bigand E. How functional coupling between the auditory cortex and the amygdala induces musical emotion: a single case study. Cortex. 2014 Nov;60:82-93. doi: 10.1016/j.cortex.2014.06.002. Epub 2014 Jun 16. PMID 25023618
- [Background] Pruvost-Robieux E, Andre-Obadia N, Marchi A, Sharshar T, Liuni M, Gavaret M, Aucouturier JJ. It's not what you say, it's how you say it: A retrospective study of the impact of prosody on own-name P300 in comatose patients. Clin Neurophysiol. 2022 Mar;135:154-161. doi: 10.1016/j.clinph.2021.12.015. Epub 2022 Jan 13. PMID 35093702
- [Background] Shestopalova LB, Petropavlovskaia EA, Semenova VV, Nikitin NI. Mismatch negativity and psychophysical detection of rising and falling intensity sounds. Biol Psychol. 2018 Mar;133:99-111. doi: 10.1016/j.biopsycho.2018.01.018. Epub 2018 Feb 5. PMID 29421188
- [Background] Goupil L, Ponsot E, Richardson D, Reyes G, Aucouturier JJ. Listeners' perceptions of the certainty and honesty of a speaker are associated with a common prosodic signature. Nat Commun. 2021 Feb 8;12(1):861. doi: 10.1038/s41467-020-20649-4. PMID 33558510